CLINICAL TRIAL: NCT04894994
Title: Phase 2 Study of FLX475 in Combination With Ipilimumab in Advanced Melanoma
Brief Title: FLX475 in Combination With Ipilimumab in Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in clinical landscape
Sponsor: RAPT Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLX475-03
Record Dates: First submitted 2021-05-12; First posted 2021-05-20 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Advanced Melanoma
Keywords: Neoplasms; Ipilimumab; Antineoplastic Agents; Immunological
MeSH Terms: conditions — Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FLX475 and ipilimumab combination therapy (Experimental): Participants received FLX475 tablets orally and ipilimumab by IV infusions
  Interventions: Drug: FLX475; Drug: Ipilimumab

INTERVENTIONS:
Drug: FLX475 — Tablet
Drug: Ipilimumab — IV infusion

SUMMARY:
This clinical trial is a Phase 2, open-label study to determine the anti-tumor activity of FLX475 in combination with ipilimumab in subjects with advanced melanoma previously treated with an anti-programmed cell death 1 (anti-PD-1) or anti-programmed cell death ligand 1 (anti-PD-L1) agent.

The study will be conducted starting with a safety run-in portion in which 6 eligible subjects will be enrolled and treated for at least one 3-week cycle to determine if the safety profile of FLX475+ipilimumab is acceptable to complete enrollment of the approximately 20-subject study.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV or unresectable Stage III advanced melanoma
* Prior treatment with at least 2 months of anti-PD-(L)1 agent
* Measurable disease at baseline
* Tumor available for biopsy

Exclusion Criteria:

* History of allergy or severe hypersensitivity to biologic agents
* History of Grade 3-4 immune-related adverse events leading to discontinuation of prior immunotherapy
* Prior treatment with ipilimumab or other (cytotoxic T-lymphocyte-associated antigen 4) CTLA-4 antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Ho, MD, PhD, Study Chair — RAPT Therapeutics, Inc.
Locations (4):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Washington University School of Medicine St. Louis, St Louis, Missouri
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FLX475 and Ipilimumab Combination Therapy
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FLX475 and Ipilimumab Combination Therapy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: To evaluate the objective response rate (ORR), defined as confirmed complete or partial response per RECIST 1.1, of FLX475 in combination with ipilimumab in subjects with advanced melanoma previously treated with an anti-PD-1 or anti-PD-L1 agent
Time Frame: Approximately 1 year
Population: This outcome was not measured as the study was prematurely terminated for reasons unrelated to safety,
Arm/Group | FLX475 and Ipilimumab Combination Therapy
Number analyzed (Participants) | 0

2. Primary Outcome: Safety and Tolerability as Measured by Number of Participants That Experienced Other Adverse Events
Description: Number of participants that experienced Other Adverse Events
Time Frame: Approximately 3 weeks
Population: Participants received FLX475 tablets orally and ipilimumab by IV infusions
Measure: Count of Participants; unit: Participants
Arm/Group | FLX475 and Ipilimumab Combination Therapy
Number analyzed (Participants) | 6
Participants | 6

3. Secondary Outcome: Progression-free Survival
Description: To evaluate the progression-free survival (PFS) of subjects with advanced melanoma treated with FLX475 in combination with ipilimumab who have been previously treated with an anti-PD-1 or anti-PD-L1 agent
Time Frame: Approximately 1 year
Population: This outcome was not measured as the study was prematurely terminated for reasons unrelated to safety.
Arm/Group | FLX475 and Ipilimumab Combination Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: To evaluate the overall survival (OS) of subjects with advanced melanoma treated with FLX475 in combination with ipilimumab who have been previously treated with an anti-PD-1 or anti-PD-L1 agent
Time Frame: Approximately 1 year
Population: All participants who received the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | FLX475 and Ipilimumab Combination Therapy
Number analyzed (Participants) | 6
Participants | 3

5. Secondary Outcome: Plasma Concentrations of FLX475
Description: To evaluate the plasma concentrations of FLX475 when it is given in combination with ipilimumab
Time Frame: Approximately 1 year
Population: This outcome was not measured as the study was prematurely terminated for reasons unrelated to safety,
Arm/Group | FLX475 and Ipilimumab Combination Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Pharmacodynamic (PD) Markers
Description: To assess the effects of FLX475 in combination with ipilimumab on pharmacodynamic (PD) markers relating to drug mechanism of action
Time Frame: Approximately 1 year
Population: This outcome was not measured as the study was prematurely terminated for reasons unrelated to safety.
Arm/Group | FLX475 and Ipilimumab Combination Therapy
Number analyzed (Participants) | 0

7. Secondary Outcome: Tumor Control
Description: To characterize the onset, magnitude, and duration of tumor control in subjects receiving FLX475 in combination with ipilimumab
Time Frame: Approximately 1 year
Population: This outcome was not measured as the study was prematurely terminated for reasons unrelated to safety.
Arm/Group | FLX475 and Ipilimumab Combination Therapy
Number analyzed (Participants) | 0

8. Primary Outcome: Safety and Tolerability as Measured by Number of Participants That Experienced Serious Adverse Events
Description: Number of participants that experienced Serious Adverse Events
Time Frame: Approximately 3 weeks
Population: Participants received FLX475 tablets orally and ipilimumab by IV infusions
Measure: Count of Participants; unit: Participants
Arm/Group | FLX475 and Ipilimumab Combination Therapy
Number analyzed (Participants) | 6
Participants | 5

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events were reported by the sites into an electronic data capture system
Arm/Group | FLX475 and Ipilimumab Combination Therapy
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLX475 and Ipilimumab Combination Therapy (N=6)
Hepatic Enzyme Increased (Investigations) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Autoimmune Colitis (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (3)
Fatigue (General disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FLX475 and Ipilimumab Combination Therapy (N=6)
Constipation (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Autoimmune colitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 4
Alanine aminotransferase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 2
Weight decreased (Investigations) | 2
Amylase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Lipase increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Autoimmune dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Taste disorder (Nervous system disorders) | 1
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 2
Chills (General disorders) | 1
Early satiety (General disorders) | 1
Influenza like illness (General disorders) | 1
Oedema peripheral (General disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic haematoma (Hepatobiliary disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
COVID-19 (Infections and infestations) | 1
Campylobacter infection (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Confusional state (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to changes in the treatment landscape of melanoma that have occurred since the initiation of the study, leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT04894994/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04894994/SAP_001.pdf